CLINICAL TRIAL: NCT06466941
Title: Impact of Patient Phenotypic Features on the Experience and Effectiveness of Regional Anesthesia and Postoperative Pain
Brief Title: Understanding the Acute Pain Phenotype in Patients Undergoing Surgery
Status: Recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Kristin Schreiber, Anesthesiologist, Brigham and Women's Hospital
Other Study IDs: 2023P003642; 2R35GM128691-06 (NIH)
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Acute Pain; Chronic Post Operative Pain; Opioid Use
Keywords: regional anesthesia; peripheral nerve blocks; psychosocial phenotype; pain catastrophizing
MeSH Terms: conditions — Acute Pain; Pain, Postoperative | interventions — Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Thoracic surgery and open abdominal surgery: Patients who underwent surgery thoracic surgery or open abdominal surgery
  Interventions: Procedure: regional anesthesia; Procedure: no regional anesthesia
- Orthopedic surgery: Patients who underwent orthopedic surgery
  Interventions: Procedure: regional anesthesia; Procedure: no regional anesthesia
- Spine surgery: Patients who underwent spine surgery
  Interventions: Other: acute pain consultation; Other: no acute pain consultation

INTERVENTIONS:
Procedure: regional anesthesia — Patients who underwent surgery and received an epidural or peripheral nerve block
  Groups: Orthopedic surgery; Thoracic surgery and open abdominal surgery
Procedure: no regional anesthesia — Patients who underwent surgery and did not received an epidural or peripheral nerve block
  Groups: Orthopedic surgery; Thoracic surgery and open abdominal surgery
Other: acute pain consultation — Patients who underwent surgery and had a perioperative (preop, intraop, or postop) acute pain consultation
  Groups: Spine surgery
Other: no acute pain consultation — Patients who underwent surgery and did not have a perioperative (preop, intraop, or postop) acute pain consultation
  Groups: Spine surgery

SUMMARY:
The goal of this observational study is to learn about how regional anesthesia (numbing medication) affects pain in patients with different psychosocial phenotypes such as different levels of concern about pain, sleep issues, and anxiety, who are having surgery.

The main questions are:

1. Do psychosocial factors such as concerns about pain, sleep, anxiety affect the effectiveness of regional anesthesia?
2. Do psychosocial factors and regional anesthesia affect the amount of opioids used after surgery?
3. Do psychosocial factors and regional anesthesia affect development of chronic postsurgical pain?

DETAILED DESCRIPTION:
A patient's psychological profile importantly modulates pain severity, and the overall experience and impact of pain. For instance, catastrophic thinking about pain, including magnification, rumination, and helplessness, is associated with both greater pain severity and impact.

Over the years, regional anesthesia has become an integral part of multimodal pain management for many surgeries. Regional anesthesia (epidural and peripheral nerve blocks) to be associated with superior pain control, reduced time to return of bowel function, shorter intraoperative times, fewer side effects and complications, earlier ambulation and functional exercise capacity post-discharge, lower in-hospital mortality, reduced length-of-stay, improved patient satisfaction, and fewer readmissions.

The investigators aim to use of validated psychosocial surveys and semi-structured interviews to understand the phenotype of patients who will benefit the most from regional anesthesia. The investigators also aim to understand how different patient phenotypes and regional anesthesia affect perioperative opioid consumption, and development of chronic postsurgical pain.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* English speaking
* Surgical or procedural patient who will be admitted postoperatively
* Willingness to answer psychosocial survey and/or audio recorded semi-structured interview

Exclusion Criteria:

-Cognitive dysfunction that precludes communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All surgical patients are eligible for the study if they meet the inclusion/exclusion criteria. We plan to enroll patients who may or may not receive a nerve block placement (ex: epidural or peripheral nerve block) during their clinical care or have a surgery that may result in an acute postoperative pain consult (ex: spine and orthopedic surgery).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Maximum pain score over the first 24 hours after surgery | 0-24 hours
  Maximum pain score (numerical pain rating score 0-10) over the first 24 hours after surgery

SECONDARY OUTCOMES:
Worst pain score over the first 24 hours after surgery | 0-24 hours
  Worst pain score (numerical pain rating score 0-10) over the first 24 hours after surgery
Average pain score over the first 24 hours after surgery | 0-24 hours
  Average pain score (numerical pain rating score 0-10) over the first 24 hours after surgery
Least pain score over the first 24 hours after surgery | 0-24 hours
  Least pain score (0-10) over the first 24 hours after surgery
Daily pain scores | 0-7days
  Comparison of pain scores (numerical pain rating score 0-10) over the first 7 days after surgery
Longitudinal pain scores | 1-12 months
  Comparison of pain scores (numerical pain rating score 0-10) at 1 month, 3 months, 6 months, and 12 months
Postoperative opioid consumption | 0-7 days
  Comparison of amount of opioids used after surgery (morphine milliequivalents)
Incidence of chronic postsurgical pain | 3-12 months
  Comparison of persistent pain in the surgical area > 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kristin L Schreiber, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen YK, Boden KA, Schreiber KL. The role of regional anaesthesia and multimodal analgesia in the prevention of chronic postoperative pain: a narrative review. Anaesthesia. 2021 Jan;76 Suppl 1(Suppl 1):8-17. doi: 10.1111/anae.15256. PMID 33426669
- [Background] Schreiber KL, Zinboonyahgoon N, Flowers KM, Hruschak V, Fields KG, Patton ME, Schwartz E, Azizoddin D, Soens M, King T, Partridge A, Pusic A, Golshan M, Edwards RR. Prediction of Persistent Pain Severity and Impact 12 Months After Breast Surgery Using Comprehensive Preoperative Assessment of Biopsychosocial Pain Modulators. Ann Surg Oncol. 2021 Sep;28(9):5015-5038. doi: 10.1245/s10434-020-09479-2. Epub 2021 Jan 15. PMID 33452600
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416